CLINICAL TRIAL: NCT01266057
Title: A Phase I Trial of Sirolimus (mTOR Inhibitor) or Vorinostat (HDAC Inhibitor) in Combination With Hydroxychloroquine (Autophagy Inhibitor) in Patients With Advanced Malignancies
Brief Title: Sirolimus or Vorinostat and Hydroxychloroquine in Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0588; NCI-2011-00303 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-12-22; First posted 2010-12-24 (Estimated); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Advanced Cancers
Keywords: Advanced Malignancies; Metastatic cancers; Sirolimus; Hydroxychloroquine; Vorinostat; Plaquenil; Rapamune; Saha; Suberoylanilide Hydroxamic Acid; MSK-390; Zolinza
MeSH Terms: conditions — Neoplasms | interventions — Hydroxychloroquine; Sirolimus; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine + Sirolimus (Experimental): Hydroxychloroquine starting dose of 200 mg by mouth every day for a 21 day cycle. Sirolimus starting dose of 2 mg by mouth every day for a 21 day cycle.
  Interventions: Drug: Hydroxychloroquine; Drug: Sirolimus
- Hydroxychloroquine + Vorinostat (Experimental): Hydroxychloroquine starting dose of 200 mg by mouth every day for a 21 day cycle. Vorinostat starting dose of 200 mg by mouth per day for a 21 day cycle.
  Interventions: Drug: Hydroxychloroquine; Drug: Vorinostat

INTERVENTIONS:
Drug: Hydroxychloroquine — Starting dose of 200 mg by mouth every day for a 21 day cycle.
  Other Names: Plaquenil
Drug: Sirolimus — Starting dose of 2 mg by mouth every day for a 21 day cycle.
  Other Names: Rapamune
  Arms: Hydroxychloroquine + Sirolimus
Drug: Vorinostat — Starting dose of 200 mg by mouth per day for a 21 day cycle.
  Other Names: SAHA; Suberoylanilide Hydroxamic Acid; MSK-390; Zolinza
  Arms: Hydroxychloroquine + Vorinostat

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of sirolimus or vorinostat that can be given in combination with hydroxychloroquine to patients with advanced cancer. The safety of these drug combinations will also be studied.

DETAILED DESCRIPTION:
Study Drug Dose Level:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of hydroxychloroquine and either sirolimus or vorinostat, based on when you joined this study, availability of spots for each drug combination, and what your doctor thinks is in your best interest. Up to 11 dose levels of the sirolimus and hydroxychloroquine combination and 7 dose levels of the vorinostat and hydroxychloroquine combination will be tested. Three (3) to 6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level of the study drug combination. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of each drug combination is found.

Once the highest tolerated dose of each drug combination is found, up to 28 more participants (14 per combination) will be given this dose. The study doctor will decide which drug combination each participant is given, based on their tumor type.

Study Drug Administration:

Each study "cycle" is 21 days.

You will take hydroxychloroquine and either vorinostat or sirolimus by mouth, 1 time a day, every day. You should take the pills at about the same time each day with food and a cup (8 ounces) of water.

Study Visits:

At every study visit, you will be asked about any health conditions you have, drugs you may be taking, and if you have had any side effects.

Weekly During Cycle 1:

° Blood (about 2 teaspoons) will be drawn for routine tests.

At the beginning of each cycle beginning with 2:

* You will have a physical exam.
* Your medical history will be recorded.
* You will be asked if you have any muscle weakness or difficulty while moving.

Every 6 weeks, you will have an x-ray, CT scan, MRI scan, and/or PET/CT to check the status of the disease. If the study doctor thinks it is needed, they will be performed more often. If you are able to become pregnant, you will have a blood (about 1 teaspoon) or urine pregnancy test.

About every 3 months, you will have an eye exam.

Length of Study:

You may continue taking the study drugs for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse or intolerable side effects occur.

This is an investigational study. Sirolimus is FDA approved and commercially available for the treatment of patients with a kidney transplant. Vorinostat is FDA approved and commercially available for the treatment of cutaneous T-cell lymphoma. Hydroxychloroquine is FDA approved and commercially available to treat malaria. The use of these drugs combinations is investigational.

Up to 224 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced or metastatic cancers that are refractory to standard therapy, relapsed after standard therapy, or who have no standard therapy available that improves survival by at least three months.
2. Patients must be >/= 18 years.
3. Patients must be >/= 3 weeks beyond treatment with a cytotoxic chemotherapy regimen, or therapeutic radiation, or major surgery. Patients may have received palliative localized radiation immediately before or during treatment provided that radiation is not delivered to the only site of disease being treated under this protocol. For biologic/targeted agents patients must be >/= 5 half-lives or >/= 3 weeks form the last dose (whichever comes first).
4. ECOG performance status </= 2
5. Patients must have adequate organ and marrow function defined as: absolute neutrophil count >/= 1,000/mL;platelets >/=50,000/mL; creatinine </= 2 X ULN; total bilirubin </= 2.0 (exceptions may apply to benign non-malignant indirect hyperbilirubinemia such as Gilbert syndrome); ALT(SGPT) </= 5 X ULN; Exception for patients with liver metastasis: total bilirubin </= 3 x ULN; ALT(SGPT) </= 8 X ULN;cholesterol </= 350 mg/dL; triglycerides </= 400 mg/dL (sirolimus and hydroxychloroquine only).
6. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 30 days after the last dose.
7. Patients must be able to understand and be willing to sign a written informed consent document.

Exclusion Criteria:

1. Uncontrolled intercurrent illness, including, but not limited to, uncontrolled infection, uncontrolled asthma, need for hemodialysis, need for ventilatory support.
2. Pregnant or lactating women.
3. History of hypersensitivity to sirolimus.
4. History of hypersensitivity to vorinostat
5. History of hypersensitivity to hydroxychloroquine
6. History of hypersensitivity to any component of the formulation.
7. Patients unwilling or unable to sign informed consent document.
8. Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.
9. Patients with known glucose-6-phosphate dehydrogenase deficiency.
10. Patients with porphyria cutanea tarda.
11. Patients with psoriasis.
12. Patients with pre-existing maculopathy or retinopathy of the eye.
13. Patients who have a pre-existing myopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2011-04-28 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Sirolimus or Vorinostat in Combination with Hydroxychloroquine in Participants with Advanced Cancers | 21 day cycles, approximately 4 weeks for DLT assessment
  Maximum tolerated dose (MTD) defined defined as the dose level below the dose at which 2 of 6 patients experience drug-related dose limiting toxicity (DLT) in the first treatment cycle.
  Dose limiting toxicity (DLT) defined as: Any grade 3 or 4 non-hematologic toxicity as defined in the NCI CTC v3.0 that is possibly, probably or definitely related to any of the three study medications, even if expected. This is to include symptoms/signs of vascular leak or cytokine release syndrome; or any severe or life-threatening complication or abnormality not defined in the NCI-CTCAE that is possibly, probably or definitely related to the therapy.

SECONDARY OUTCOMES:
Antitumor Efficacy of Sirolimus or Vorinostat in Combination with Hydroxychloroquine in Participants with Advanced Cancers | 6 weeks
  Participants with lymphoma measured per the WHO criteria,68 and all others evaluated using RECIST 1.1 criteria.69.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Janku, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org